CLINICAL TRIAL: NCT03339362
Title: A Multicentre Double-blind Randomised Controlled Trial to Assess the Clinical- and Cost-effectiveness of Facet-joint Injections in Selected Patients With Non-specific Low Back Pain: a Feasibility Study
Brief Title: FAcet-joint Injection Clinical and Cost-effective Trial
Acronym: FACET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Facet-joint feasibility study
Record Dates: First submitted 2014-09-01; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-06

CONDITIONS: Low Back Pain
Keywords: low back pain; lumbar facet joint pain; feasibility; lumbar facet joint injection
MeSH Terms: conditions — Low Back Pain | interventions — Bupivacaine; Methylprednisolone; Methylprednisolone Acetate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients with persistent low back pain, referred to a community or hospital-based pain clinic by their general practitioner, will be reviewed and assessed by a pain physiotherapist and pain physician. They will be screened and recruited based on clinical history and examination. Participants will receive diagnostic injections (medial branch nerve blocks); those with a positive response will randomly receive either steroid FJIs or a sham procedure, under x-ray guidance.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Procedure (Active Comparator): All patients will receive 6 X-ray guided peri-articular injections via a spinal needle at 2 bilateral lumbar levels using 0.5ml of 1% Lidocaine. This a test procedure to identify the patient has a 50% pain reduction from baseline pain numerical score. If patients pass this test injection, they will be randomised to the active or sham procedure.
  4 X-ray guided intra-articular facet-joint injections via a spinal needle at 2 bilateral lumbar levels, using 0.5ml 0.5% bupivacaine + 20mg methylprednisolone per joint
  Interventions: Procedure: Active Procedure
- Sham procedure (Sham Comparator): All patients will receive 6 X-ray guided peri-articular injections via a spinal needle at 2 bilateral lumbar levels using 0.5ml of 1% Lidocaine. This a test procedure to identify the patient has a 50% pain reduction from baseline pain numerical score. If patients pass this test injection, they will be randomised to the active or sham procedure.
  4 X-ray guided peri-articular injections via a spinal needle at 2 bilateral lumbar levels using 0.5ml normal saline per injection
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Active Procedure — If they pass the diagnostic injection with a 50% or more in pain reduction, they are randomised to receive either the active procedure or sham procedure.
  Active: 4 X-ray guided intra-articular lumbar facet-joint injections via a spinal needle at 2 bilateral lumbar levels using 0.5ml bupivacaine + 20mg methylprednisolone per joint
  Other Names: Active group; 0.5% bupivacaine + 20mg methylprednisolone; Depo-medrone + Bupivacaine
  Arms: Active Procedure
Procedure: Sham procedure — If they pass the diagnostic injection with a 50% or more in pain reduction, they are randomised to receive either the active procedure or sham procedure.
  Sham: 4 X-ray guided peri-articular injections via a spinal needle at 2 bilateral lumbar levels using 0.5ml of 0.9% sodium chloride per joint.
  Other Names: Sham group; 0.9% sodium chloride; normal saline; placebo
  Arms: Sham procedure

SUMMARY:
Lumbar facet-joints are small, paired joints in the low back that provide stability, integrity and flexibility of movement to the spine. Diseased facet-joints may cause persistent low back pain, with significant socioeconomic impact. At present, there is insufficient high quality evidence to support the use of lumbar facet-joint injections (FJIs) in treating low back pain of less than 12 months' duration; the National Institute for Health and Care Excellence (NICE) therefore did not approved their use in their 2009 publication.

This study will investigate the feasibility of conducting a larger, definitive trial to assess lumbar FJIs (a needle is inserted into the facet-joint and steroid injected), by comparing it to a dummy or 'sham' procedure (a needle is inserted near the facet-joint but no therapeutic substance injected).

Patients with persistent low back pain, referred to a community or hospital-based pain, spinal or musculoskeletal clinic by their general practitioner, will be reviewed and assessed by a specialist physician. They will be screened and recruited based on clinical history and examination. Participants will receive diagnostic injections (medial branch nerve blocks); those with a positive response will randomly receive either FJIs or a sham procedure, under x-ray guidance. All participants will receive a combined physical and psychological programme recommended by NICE as a strategy to reduce pain and its impact on the person's day-to-day life, even if the pain cannot be cured completely.

Participants will be asked to complete questionnaires comparing a range of pain and disability-related issues. These will occur at baseline (before treatment) and at 6 weeks, 3 months and 6 months after their injections.

Criteria for the study to be considered successful (and a definitive trial feasible) include the abilities to standardise the methods for injection and to recruit and retain sufficient participants, and the acceptability of the study design to participants and clinicians.

DETAILED DESCRIPTION:
Design

This study seeks to examine the feasibility of undertaking a fully powered double-blind randomised controlled trial. Patients with non-specific low back pain of more than three months' duration with confirmed facet-joint disease will be individually randomised 1:1 to receive facet-joint injections plus a combined physical and psychological programme (intervention group) or to a sham (placebo) procedure plus a combined physical and psychological programme (control group).

Setting

The feasibility study will be conducted in three hospital-based pain medicine centres: Barts Health NHS Trust (formerly Barts and The London NHS Trust), Basildon and Thurrock University Hospitals NHS Foundation Trust, and The Walton Centre NHS Foundation Trust.

Target population

Patients will be recruited from pain, spinal and musculoskeletal clinics at the three participating NHS centres and their associated community clinics. Patients will be referred by their general practitioners with low back pain requiring further specialist assessment, for reasons such as uncertain diagnosis, failure of conservative treatment, or expectation of therapeutic interventions. A screening visit will be used to identify eligible patients i.e. pain of at least 3 months' duration and an average pain intensity numerical rating score (NRS) of at least 4/10 in the 7 preceding days, signs and symptoms of facet-joint disease including bilateral localised paraspinal tenderness at 2 lumbar levels, and have received two components of NICE-defined best non-invasive care (education and one of: physical exercise programme, acupuncture, or manual therapy).

Health technologies being assessed

Facet-joint injections of local anaesthetic and steroid for non-specific low back pain. (Delivered in this study as four X-ray guided intra-articular facet-joint injections through a spinal needle at two lumbar levels bilaterally, using 0.5ml 0.5% bupivacaine + 20mg methylprednisolone per joint, under fluoroscopic guidance.)

Measurement of costs and outcomes

The primary outcomes for this feasibility study include: patient recruitment and attrition rates, levels of patient completion of outcomes, acceptability of the study design to patients and clinicians, fidelity of sham injection and process of blinding, and collection of variance outcome data to inform a future sample size calculation.

The investigators have proposed stopping rules for progression to a main trial. The proposed outcomes for the main trial have been selected in accord with IMMPACT recommendations for chronic pain trials and include: pain assessment, psychological well-being, health-related quality of life, functional disability, health care utilisation including analgesic usage, lost productivity and complications/level of adverse events. Outcomes will be collected at clinic visits at baseline (pre-randomisation) and at 6 weeks, 3 months, and 6 months post-randomisation.

Sample size

The investigators will recruit a total of 150 patients who will undergo a diagnostic facet-joint injection to determine eligibility to participate (test positive for facet-joint disease). Sixty participants (40% of all recruited) are expected to have a positive response to the diagnostic test; these 60 patients will be randomly and equally allocated to intervention and control groups. Assuming up to a 33% attrition rate, the investigators will have >24 complete data sets per arm at the end of the study. This sample size will allow us to achieve our various feasibility objectives.

Project timetables including recruitment rate

A retrospective audit of patient throughput in participating clinics shows that recruitment to achieve 30 patients per treatment arm is readily feasible in the time frame of this study. From 1000 new patient attendances for low back pain at the pain services, the investigators expect approximately 1 in 4 patients to be eligible to enter the study. This is based on our clinical experience and published studies based on responses to controlled diagnostic facet-joint injections, performed in accordance with the criteria established by the International Association for the Study of Pain. Of these 250 patients, approximately 60% (150) will consent to enter the study, of whom approximately 40% (60 patients) are expected to have a positive response from diagnostic medial branch nerve blocks.

The investigators anticipate that the project will take a total of 21 months to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70 years attending pain clinics identified during routine clinical assessment of non-specific low back pain (clinical indicators for pain of facet-joint origin include tenderness over the facet-joints, referred leg pain above the knees, and worsening pain on extension, flexion and rotation).
2. Low back pain of greater than three months' duration.
3. Average pain intensity score of 4/10 or more in the seven days preceding recruitment despite NICE-recommended treatment (NICE recommends providing patients with advice and information to promote self-management of their low back pain, and offering one of the following treatments, taking into account patient preference: an exercise programme, a course of manual therapy, or a course of acupuncture).
4. Dominantly paraspinal (not midline) tenderness at two bilateral lumbar levels.
5. At least two components of NICE-recommended best non-invasive care completed, including education and one of a physical exercise programme, acupuncture, and manual therapy.

Exclusion Criteria:

1. Patient refusal.
2. More than four painful lumbar facet-joints.
3. Patient has not completed at least two components of NICE-recommended best non-invasive care.
4. 'Red flag' signs ('Red flag' signs are possible indicators of serious spinal pathology, and include thoracic pain, fever, unexplained weight loss, bladder or bowel dysfunction, progressive neurological deficit, and saddle anaesthesia).
5. Hypersensitivity to study medications or X-ray contrast medium.
6. Radicular pain (Radicular pain is defined as pain perceived as arising in a limb or the trunk wall caused by ectopic activation of nociceptive afferent fibres in a spinal nerve or its roots or other neuropathic mechanisms. The pain is lancinating in quality and travels along a narrow band).
7. Dominantly midline tenderness over the lumbar spine.
8. Any other dominant pain.
9. Any major systemic disease or mental health illness that may affect the patient's pain, disability and/or their ability to exercise and rehabilitate.
10. Any active neoplastic disease, including primary or secondary neoplasm.
11. Pregnant or breastfeeding patients.
12. Previous lumbar facet-joint injections.
13. Previous lumbar spinal surgery.
14. Patients with morbid obesity (body mass index of 35 or greater).
15. Major trauma or infection to the lumbar spine.
16. Participation in another clinical trial in the past thirty days.
17. Patients unable to commit to the six-month study duration.
18. Patients involved in legal actions or employment or benefit tribunals related to their low back pain.
19. Patients with a history of substance abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Pain numerical rating scale (NRS) | Baseline (visit 1) and diagnostic injections (visit 2)
  The rationale for carrying out diagnostic medial branch nerve blocks is because of their safety, simplicity and prognostic value.
  There is currently no justification for double, comparative blocks as these are associated with a significant false-negative rate and are not shown to be cost-effective.
  The pain scores at baseline (recruitment) will be recorded using a numerical rating scale (0-10) and will be compared to the score taken 20-40 minutes and 180-200 minutes after the injections. If a positive response of 50% pain reduction is seen, we know the pain is definately coming from the facet- joint which entitles the patient to be eligible for the randomised procedure.

SECONDARY OUTCOMES:
Change in Pain intensity and characteristics: Brief Pain Inventory (BPI) (Short Form) Modified, with its 11-point NRS Short Form McGill Pain Questionnaire. | Baseline (visit 1)
  Pain assessments to assess change in outcome measure in the form of questionnaires.
Change in Pain intensity and characteristics: Brief Pain Inventory (BPI) (Short Form) Modified, with its 11-point NRS Short Form McGill Pain Questionnaire. | 6 weeks (visit 4)
  Pain assessments to assess change in outcome measure in the form of questionnaires. This will be compared with responses from the baseline visit.
Change in Pain intensity and characteristics: Brief Pain Inventory (BPI) (Short Form) Modified, with its 11-point NRS Short Form McGill Pain Questionnaire. | 3 months (visit 5)
  Pain assessments to assess change in outcome measure in the form of questionnaires. This will be compared with responses from the baseline visit.
Change in Pain intensity and characteristics: Brief Pain Inventory (BPI) (Short Form) Modified, with its 11-point NRS Short Form McGill Pain Questionnaire. | 6 months (visit 6)
  Pain assessments to assess change in outcome measure in the form of questionnaires. This will be compared with responses from the baseline visit.
Expectation of benefit | Baseline
  0 to 6 scale, ranging from "expect no improvement" to "expect total improvement".
Change in Health-related quality of life: EQ5D-5L, 12-item Short Form Survey (SF-12) at different follow- up visits | Baseline (visit 1), 6 weeks (visit 4), 3 months (visit 5) and 6 months (visit 6)
  Pain assessments to assess change in outcome measure in the form of questionnaires.
Change in Functional impairment: Oswestry Low Back Pain Disability Questionnaire, Pain Self Efficacy Questionnaire (PSEQ) at different follow-up visits | Baseline (visit 1)
  Pain assessments to assess change in outcome measure in the form of questionnaires.
Change in Co-psychological well-being: Hospital Anxiety and Depression Scale, Pain Catastrophizing Scale, SF-12, BPI at different follow up visits | 6 weeks (visit 4)
  Pain assessments to assess change in outcome measure in the form of questionnaires.This will be compared with responses from the baseline visit.
Change in Co-psychological well-being: Hospital Anxiety and Depression Scale, Pain Catastrophizing Scale, SF-12, BPI at different follow up visits | 3 months (visit 5)
  Pain assessments to assess change in outcome measure in the form of questionnaires.This will be compared with responses from the baseline visit.
Change in Co-psychological well-being: Hospital Anxiety and Depression Scale, Pain Catastrophizing Scale, SF-12, BPI at different follow up visits | 6 months (visit 6)
  Pain assessments to assess change in outcome measure in the form of questionnaires.This will be compared with responses from the baseline visit.
Change in Healthcare utilisation and costs, and impact on productivity at different follow up visits | Baseline (visit 1)
  This will include the use if published national costs to calculate costs of delivering each treatment arm/intervention and downstream healthcare utilization. The tools to assess this are the Stanford Presenteeism Scale 6, self-reported measures of sickness absence over the previous 3 months, and healthcare utilisation in the form of hospital visits, treatments and medications.
Change in Healthcare utilisation and costs, and impact on productivity at different follow up visits | 6 weeks (visit 4)
  This will include the use if published national costs to calculate costs of delivering each treatment arm/intervention and downstream healthcare utilization. The tools to assess this are the Stanford Presenteeism Scale 6, self-reported measures of sickness absence over the previous 3 months, and healthcare utilisation in the form of hospital visits, treatments and medications.This will be compared with responses from the baseline visit.
Change in Healthcare utilisation and costs, and impact on productivity at different follow up visits | 3 months (visit 5)
  This will include the use if published national costs to calculate costs of delivering each treatment arm/intervention and downstream healthcare utilization. The tools to assess this are the Stanford Presenteeism Scale 6, self-reported measures of sickness absence over the previous 3 months, and healthcare utilisation in the form of hospital visits, treatments and medications.This will be compared with responses from the baseline visit.
Change in Healthcare utilisation and costs, and impact on productivity at different follow up visits | 6 months (visit 6)
  This will include the use if published national costs to calculate costs of delivering each treatment arm/intervention and downstream healthcare utilization. The tools to assess this are the Stanford Presenteeism Scale 6, self-reported measures of sickness absence over the previous 3 months, and healthcare utilisation in the form of hospital visits, treatments and medications.This will be compared with responses from the baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Mehta, MBBS, Study Director — Barts & The London NHS Trust
Locations (3):
- United Kingdom (3):
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon, Essex
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
No plans are made to share individual participant data